CLINICAL TRIAL: NCT02783118
Title: Using a Smartphone App to Reduce Cognitive Vulnerability and Mild Depressive Symptoms: An Exploratory Study Protocol for a Randomized Controlled Trial
Brief Title: Using a Smartphone App to Reduce Cognitive Vulnerability and Mild Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Cezar Giosan, PhD, Principal Investigator, PhD, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EEA-JRP-RO-NO-2013-1-0358/1
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Mild Depression
Keywords: Depression; Prevention; CBT; Smartphone app
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy sample, active intervention (Experimental): Healthy participants will be testing a depression prevention app employing a self administered online CBT intervention, for 4 weeks.
  Interventions: Other: Self administered online CBT
- Healthy sample, delayed intervention (No Intervention): Healthy participants will be put on a wait list for 4 weeks, after which access to the depression prevention app will be given.
- Mild depression, active intervention (Experimental): Mildly depressed participants will be testing a depression prevention app, employing a self administered online CBT intervention, for 4 weeks.
  Interventions: Other: Self administered online CBT
- Mild depression, delayed intervention (No Intervention): Mildly depressed participants will be put on a wait list for 4 weeks, after which access to the depression prevention app will be given.

INTERVENTIONS:
Other: Self administered online CBT — The app being tested has two main components: courses and exercises. Courses represent the psycho-educational and therapeutic background of the program, comprising the following topics: information on depression, psychological vulnerability, what is CBT, healthy and unhealthy negative emotions, rational and irrational thoughts, how behaviors contribute to depression, sleep hygiene, social support, and relaxation techniques. Exercises use the information presented in the courses and follow the structure of a regular therapy session and/or therapeutic homework.
  The following exercises are included in the app:
  1. The Emotional Pulse exercise
  2. The Sticky Notes exercise
  3. The Find Irrational Thoughts
  4. The Change Irrational Thoughts
  Arms: Healthy sample, active intervention; Mild depression, active intervention

SUMMARY:
Depression is one of the major challenges worldwide, with significant increasing personal, economic, and societal costs. Although empirically supported treatments have been developed, they are not always available for patients in routine clinical care. Even when patients are adequately treated, they do not always respond to treatment and/or face a significant risk for recurrence. Therefore, effective and wide accessible strategies to prevent the onset of the very first depressive symptoms are necessary. Mental health apps could prove a valuable alternative for that. Although preliminary research has indicated that apps could be useful in treating depression, no study has attempted to test their utility in preventing depression symptoms. The current study aims to contrast the efficacy of a smartphone app in preventing depression compared against a waiting list condition. The app includes self-help materials and exercises based on cognitive behavioral therapy (CBT) for depression, presented in a tailored manner and incorporating gamification elements aimed at boosting the motivation to use the app.

This study protocol is the first that capitalizes on the ubiquity of smartphones to large-scale dissemination of CBT-based strategies aimed at preventing depression in nonclinical populations. The objective of this study is to test an app designed to decrease general cognitive vulnerability and promote engagement in protective, adaptive activities, while counteracting the tendency of premature dropout (through gamification and customization).

DETAILED DESCRIPTION:
Trials design. This study will include two parallel-randomized trials, with pre-post measurements. The designs of the trials will be similar and compliant with the CONSORT guidelines. In the first trial the efficacy of the preventative version of the application will be tested against a wait list control group, in a healthy sample of participants. In the second trial the efficacy of the app will be tested against a wait list control group, in a sample of participants with mild depressive symptoms.

Participant timeline. Potential participants will be assessed for eligibility through an initial assessment of depressive symptoms. The initial assessment phase consists of administration of the PHQ-9 and a short screening telephone interview. Subsequent assessments consist of all the instruments presented in the Outcome measures section. After the initial assessment, the participants meeting inclusion criteria will be randomly assigned to one of the two conditions: immediate online intervention condition (Group 1) or the delayed-intervention condition (wait-list) (Group 2).

Participants assigned to Group 1 will be given access to the online application along with explicit instructions regarding the use of all of its sections. Participants will be given 4 weeks to complete the intervention, during which time weekly messages will be sent out to them. Messages include regular assignments designed for a complete and thorough use of the application's courses and exercises, and encourage the review of materials whenever possible. However, participants are free to use the application at their own pace.

Participants in the delayed intervention group (Group 2) are placed on a wait-list for 4 weeks.

Sample size. A a total number of 50 participants per study (i.e., 50 participants without depressive symptomatology, and 50 participants with mild depressive symptomatology) was estimated based on previous studies testing mobile phone applications for depression that reported large within group effect sizes. The calculation of the sample size was conducted with G*Power 3.1. for ANOVA (Repeated measures, between factors), assuming an alpha level of 0.05, a statistical power of 0.80, and a large effect size (Cohen's f = 0.355).

Recruitment. Possible participants are approached through presentations at various events and ads in the media. Those interested in using the application are asked to provide their contact details and are subsequently contacted via e-mail, at which point the enrollment procedure is described. Initially, possible participants are invited to access the study's website and, after carefully reading the information package and informed consent, instructions to create an online account are given. The participants are then asked to answer a few demographic questions and complete the PHQ-9, to determine their eligibility for further evaluation. If eligible, a screening procedure is implemented. A short telephone interview screens out individuals whose participation in the study is motivated by problems other than their mood. Applicants who do not meet the inclusion criteria are informed via e-mail, thanked for their interest, given a summary score and interpretation for their PHQ-9 score. Applicants are encouraged to discuss their problems with a professional, if necessary. Information on how to reach one - a clinical psychologist or psychotherapist - is also provided. Licensed, certified clinical psychologists recruit prospective participants into the study. Media avenues (e.g., social networks, dedicated websites) are used for recruitment purposes. Additionally, clinicians from the private practice area are contacted for referrals.

Assignment to study group. The participants are assigned to one of the two trials, depending on their depressive symptomatology level (i.e., PHQ-9 score). Using the software Randomizer.org, participants are then randomly distributed to one of the trials' conditions. Randomization is performed by a research assistant using a simple (unrestricted) randomization sequence that assigns two unique numbers per participant; the number assigned is either 1 or 2, according to the number of the experimental conditions. To conceal the allocation mechanism, the same research assistant will monitor the assessments and allow access to the application for the participants in the delayed intervention condition (Group 2), after 1 month. The principal investigator and the statisticians running the data analysis will remain blinded to the study condition until the completion of the study.

Monitoring study implementation. Two clinical psychologists, members of the study team, screen for the risk of unintended effects or harm to the participants (i.e., clinically significant increase in depressive symptomatology, as measured by the CESD-R). The psychologists also monitor the weekly online evaluations and clinically interpret the CESD-R score of every participant. If the participant does not complete the CESD-R evaluation, a telephonic contact follows. If necessary, the supervisor can decide to interrupt the participant's access to the application and make a further referral.

ELIGIBILITY:
Inclusion Criteria:

* Romanian-speaking adults (18 years or older)
* Access to a computer, a smartphone (Android or iOS) and Internet
* A Patient Health Questionnaire-9 (PHQ-9) score of 4 or below (for the healthy participants sample)
* A PHQ-9 score no greater than 9 (for the mildly depressed participants sample)

Exclusion Criteria:

* Undergoing therapy
* Substance abuse problems
* Psychotic symptoms
* Organic brain disorders (e.g., dementia)
* Self-injury or harming others
* Serious legal or health issues that would prevent from using the app
* Reporting scores larger than 1 to Question 9 (suicidal ideation) on the (PHQ-9)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) (change from baseline) | Baseline, 1 week after baseline, 2 weeks after baseline, 3 weeks after baseline, post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  The CESD-R is a 20-item self-report instrument, which measures symptoms of depression in nine different groups: sadness (dysphoria), loss of interest (anhedonia), appetite, sleep, thinking/concentration, guilt (worthlessness), tired (fatigue), movement (agitation), and suicidal ideation. Participants rate each item on a five-point Likert scale, from 0 (not at all or less than one day) to 4 (nearly every day for 2 weeks) and refer to a time frame of a week or so. The Total CESD-R Score is calculated as a sum of responses to all 20 questions. The CESD-R exhibited good psychometric properties, including high internal consistency, strong factor loadings, and theoretically consistent convergent and divergent validity with anxiety, schizotypy, and positive and negative affect. CESD-R has been adapted to Romanian for the purposes of the current study.
The Dysfunctional Attitudes Scale Short Form (DAS-SF) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  DAS was designed to measure the intensity of dysfunctional attitudes that, according to the cognitive theory of depression, contribute to vulnerability for depression. For the purpose of this study, the short form of this scale was used. The Dysfunctional Attitudes Scale-Short Form (DAS-SF) consists of two subscales: "dependency" (6 items) and "perfectionism/performance evaluation" (11 items). The 17 items are rated on a seven-point Likert scale, from 1 (total disagreement) to 7 (total agreement). DAS-SF possesses good psychometric properties in terms of model fit, reliability and convergent construct validity. DAS-SF has been adapted to Romanian for the purposes of this study.
The Beliefs Scale (BS) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  The Beliefs Scale (BS) measures irrational beliefs. It consists of 20 items and responders indicate the level of agreement/disagreement with each item using a five-point Likert scale that ranges from 1 (strongly disagree) to 5 (strongly agree). The BS shows good psychometric properties regarding construct and discriminant validity. This scale has been translated into Romanian for the purposes of this study.
The Automatic Thoughts Questionnaire (ATQ) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  The Automatic Thoughts Questionnaire (ATQ) is a 15-item self-report measure used to assess depression-related cognitions. Participants rate, on a five-point Likert scale from 1 (never) to 5 (almost all the time), the frequency of a given thought over the past week. A higher score shows a higher frequency of automatic thoughts. The psychometric properties of the ATQ have been adequately demonstrated in previous studies. The ATQ has been successfully used on the Romanian population before.

SECONDARY OUTCOMES:
The Positive and Negative Affect Scale (PANAS) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  The Positive and Negative Affect Scale (PANAS) is a 20-item self-report questionnaire designed to assess mood. It consists of 10 items that address positive affect (PA) and 10 items that address negative affect (NA). Participants rate each item on a five-point Likert scale, from 1 (very slightly/not at all) to 5 (extremely). The PANAS can be used to assess mood on various time scales by altering the instructions. For the purposes of this study a two-week timeframe has been used. The validity and internal consistency of the PANAS are good, with test-retest reliability being the highest for the "general" temporal instruction. The PANAS has been used previously on the Romanian population and was found to have adequate psychometric properties.
Satisfaction with Life (SWL) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  Satisfaction with Life (SWL) is a five-item scale designed to measure global cognitive judgments of one's life satisfaction. Participants rate each of the 5 items using a seven-point scale that ranges from 7 (strongly agree) to 1 (strongly disagree). The SWL has been shown to be a valid and reliable measure of life satisfaction, which can be used with a wide range of age groups. SWL has been adapted to Romanian for the purposes of the current study.

OTHER OUTCOMES:
The Behavioural Activation for Depression Scale - Short Form (BADS-SF) (change from baseline) | Baseline, mid-intervention (2 weeks after baseline), post-intervention (4 weeks after baseline), Follow-up 1 (3 months after post-interv.), Follow-up 2 (6 months after post-interv.), Follow-up 3 (12 months after post-interv.)
  The Behavioural Activation for Depression Scale - Short Form (BADS-SF) is an instrument designed to be administered weekly to measure changes in avoidance and activation over the course of the Behavioral Activation (BA) treatment for depression. The BADS consists of 9 items grouped into two subscales (Activation and Avoidance/Rumination). Respondents rate each item on a seven-point Likert scale ranging from 0 (not at all) to 6 (completely). The scale enjoys good psychometric properties. BADS-SF has been translated into Romanian for the purposes of this study.
Satisfaction with the Application Scale | Post-intervention (4 weeks after baseline)
  Satisfaction with the Application Scale was specifically designed for this study. It consists of 10 items that assess users' satisfaction with the application, its difficulty level, attractiveness, and subjective utility. The first 8 items are rated on a three-point scale, ranging from 0 to 2. Each response scale is personalized to the content of the item (e.g., How attractive did you find the exercises included in the application? - 0 = rather unattractive, 1 = attractive enough; 2 = very attractive). Item 9 assesses the application globally, with the participant being asked to give an overall grade between 1 (minimum) and 10 (maximum). Item 10 asks the participants if they would recommend the application to a friend ("yes" or "no" answer).
The Application Use Scale (change from baseline) | 1 week after baseline, 2 weeks after baseline, 3 weeks after baseline, 4 weeks after baseline
  The Application Use Scale was also developed specifically for this study. It consists of 8 items that assess weekly quantitative app usage aspects: the effort invested in homework (1 item), number of practiced exercises (1 item), number of read courses (1 item), frequency of general application use (1 item), and frequency of every exercise use (4 items).

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cuijpers P, Beekman AT, Reynolds CF 3rd. Preventing depression: a global priority. JAMA. 2012 Mar 14;307(10):1033-4. doi: 10.1001/jama.2012.271. No abstract available. PMID 22416097
- [Background] Munoz RF, Beardslee WR, Leykin Y. Major depression can be prevented. Am Psychol. 2012 May-Jun;67(4):285-95. doi: 10.1037/a0027666. PMID 22583342
- [Background] Buntrock C, Ebert DD, Lehr D, Smit F, Riper H, Berking M, Cuijpers P. Effect of a Web-Based Guided Self-help Intervention for Prevention of Major Depression in Adults With Subthreshold Depression: A Randomized Clinical Trial. JAMA. 2016 May 3;315(17):1854-63. doi: 10.1001/jama.2016.4326. PMID 27139058
- [Background] Birney AJ, Gunn R, Russell JK, Ary DV. MoodHacker Mobile Web App With Email for Adults to Self-Manage Mild-to-Moderate Depression: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2016 Jan 26;4(1):e8. doi: 10.2196/mhealth.4231. PMID 26813737
- [Derived] Giosan C, Mogoase C, Cobeanu O, Szentagotai Tatar A, Muresan V, Boian R. Using a smartphone app to reduce cognitive vulnerability and mild depressive symptoms: Study protocol of an exploratory randomized controlled trial. Trials. 2016 Dec 28;17(1):609. doi: 10.1186/s13063-016-1740-3. PMID 28031038